CLINICAL TRIAL: NCT04984824
Title: Comparing the Effects of 10, 30 and 60 Minute Naps on Cognitive Performance and Memory Encoding
Brief Title: Effects of Varying Duration of Naps on Cognitive Performance and Memory Encoding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Michael WL Chee, MBBS, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NapTitration
Record Dates: First submitted 2021-03-15; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No nap group (No Intervention): No nap opportunity will be given in this condition.
- 10 minute nap (Experimental): Participants will be given a 10 minute nap.
  Interventions: Behavioral: Nap duration
- 30 minute nap (Experimental): Participants will be given a 30 minute nap.
  Interventions: Behavioral: Nap duration
- 60 minute nap (Experimental): Participants will be given a 60 minute nap.
  Interventions: Behavioral: Nap duration

INTERVENTIONS:
Behavioral: Nap duration — A cognitive battery which will be repeated at 1505, 1530, 1600 and 1900. Material for the picture encoding task will be learned at 1630 and will be tested at 2000.
  Arms: 10 minute nap; 30 minute nap; 60 minute nap

SUMMARY:
To evaluate the nap duration that achieves maximal cognitive gain with practicality of implementation, the present work employs a within-subject design comparing nap durations of 10 minutes, 30 minutes, and 60 minutes with a no nap condition on benefits to alertness, vigilance, mood, speed of processing and memory over post-nap intervals of 5 minutes, 30 minutes, 60 minutes and 240 minutes. The effect of nap duration on memory encoding will also be examined.

DETAILED DESCRIPTION:
Naps are a global phenomenon and a commonly adopted lifestyle countermeasure to reduce sleepiness and performance impairments. Experimental studies have also shown that naps can improve cognitive functioning and enhance memory and mood. However, the implementation of naps is highly varied amongst individuals, and it remains uncertain what duration of naps achieves the greatest cognitive benefit. Given the potential for naps to boost productivity in societies such as ours where insufficient nocturnal sleep is prevalent and where work hours are long, an investigation of the optimal nap duration is warranted.

Previous studies suggest that the benefits of brief naps (5-15 minutes) occur immediately after the nap and last a limited period (1-3 hours). Longer naps (>30 minutes) are more likely to produce some temporary decrements due to sleep inertia but have the potential to improve cognitive performance for a more sustained period. These findings need to be strengthened through replication and extended to include memory measures that are evaluated over a longer post-nap testing period. To evaluate the nap duration that achieves maximal cognitive gain with practicality of implementation, the present work employs a within-subject design comparing nap durations of 10 minutes, 30 minutes, and 60 minutes with a no nap condition on benefits to alertness, vigilance, mood, speed of processing and memory over post-nap intervals of 5 minutes, 30 minutes, 60 minutes and 240 minutes. The effect of nap duration on memory encoding will also be examined.

The investigator's findings are expected to inform theoretical models of sleep and cognition and will aid in the design of practical lifestyle strategies to alleviate sleepiness and improve cognitive performance that may be adopted in an everyday context to boost societal well-being and productivity.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged from 21 - 35 years and who have an average sleep duration of 6-6.5 h are eligible for this study.

Exclusion Criteria:

* Participants who have an average sleep duration of less than 6 h or more than 6.5 h, who report sleep apnea symptoms, who report drinking more than 5 cups of caffeinated drinks a day, who have a BMI greater or equal to 30, or report elevated depression or anxiety symptoms will be excluded.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Picture encoding task | In total: 35-45 min
  Participants will observe pictures of non-famous people, landscapes, scenes and objects. Later they are tested on whether they remember seeing the picture previously or not. The encoding session will take 20-30 min, and the retrieval session will take 15 min.
Levels of sleepiness | 1 min
  Karolinska Sleepiness Scale. Participants rated their level of subjective sleepiness on a 9-point Likert scale (1 - very alert, 9 - very sleepy, great effort to keep awake).
Mood | 1 min
  Positive and Negative Affect Scale. On the Positive and Negative Affect Scale (PANAS), participants responded to 20 adjectives describing positive and negative mood states on a 5-point Likert scale (1 - very slightly, 5 - extremely). Positive and negative affect scores are represented by the sum of the item responses.
Vigilance | 3 min
  Psychomotor Vigilance Test. The 3-min PVT assessed levels of sustained attention. At intervals varying randomly from 2000 ms to 10000 ms, a counter on the screen appeared and participants were to press a key as quickly as possible. Lapses were defined as responses exceeding 500 ms.
Speed of processing | 2 min
  Digit Symbol Substitution Test. The 2-min DSST was used as a measure of speed of processing. In this task, participants were required to match symbols to digits as quickly as possible following a key shown on screen. The total number of correct trials was used as the critical measure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chee, MBBS, Principal Investigator — National University of Singapore
Locations (1):
- Yong Loo Lin School of Medicine, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leong RLF, Lau T, Dicom AR, Teo TB, Ong JL, Chee MWL. Influence of mid-afternoon nap duration and sleep parameters on memory encoding, mood, processing speed, and vigilance. Sleep. 2023 Apr 12;46(4):zsad025. doi: 10.1093/sleep/zsad025. PMID 36775965